CLINICAL TRIAL: NCT04679584
Title: COVIDOM: Longterm Morbidity of SARS-CoV-2 Infection and COVID-19 Disease - Consequences for Health Status and Quality of Life (NAPKON-POP)
Brief Title: COVIDOM: Longterm Morbidity of SARS-CoV-2 Infection and COVID-19 Disease - Consequences for Health Status and Quality of Life
Acronym: NAPKON-POP
Status: Recruiting | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: Charite University, Berlin, Germany (Other); Wuerzburg University Hospital (Other); German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor
Other Study IDs: COVIDOM-Protokoll_V01F_2020-10; DRKS00023742 (Other: Deutsches Register Klinischer Studien (German Registry for Clinical Studies))
Record Dates: First submitted 2020-12-16; First posted 2020-12-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; COVID-19; COVID; Corona; longterm morbidity; Quality of Life; longterm consequences; Chronic impairment; Chronic dysfunction; Chronicity; Sequels
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Populationbased Platform (POP) of the National Pandemic Cohort Network (NAPKON): Streamlined sampling of biomaterials and core data elements (GErman Corona COnsensu data set, GECCO) with other NAPKON study platforms (HAP, SUEP).
  Interventions: Other: Observation of different courses of SARS-CoV-2 infection in different phases (acute vs. post-acute) and settings
- High-Resolution Platform (HAP) of the National Pandemic Cohort Network (NAPKON): Streamlined sampling of biomaterials and core data elements (GErman Corona COnsensu data set, GECCO) with other NAPKON study platforms (POP, SUEP).
  Interventions: Other: Observation of different courses of SARS-CoV-2 infection in different phases (acute vs. post-acute) and settings
- Intersectoral Platform (SUEP) of the National Pandemic Cohort Network (NAPKON): Streamlined sampling of biomaterials and core data elements (GErman Corona COnsensu data set, GECCO) with other NAPKON study platforms (HAP, POP).
  Interventions: Other: Observation of different courses of SARS-CoV-2 infection in different phases (acute vs. post-acute) and settings

INTERVENTIONS:
Other: Observation of different courses of SARS-CoV-2 infection in different phases (acute vs. post-acute) and settings — Oberservatory Cohorts focusing (I) on subjects after SARS-CoV-2 infection that are recruited from the general population (POP), and on subjects with acute SARS-CoV-2 infections recruited (II) in university hospital high-care settings or (III) general health care

SUMMARY:
COVID-19 is a novel disease caused by SARS-CoV-2 that primarily affects the lungs but also various other organs of the body already in early stages of the disease. Due to the multiple organ involvements in the acute phase, it is conceivable that - in a significant proportion of patients - longterm sequels in various organ systems might occur, thereby impacting the individual's health status and quality of life; and posing a relevant burden to the resources of the health care system

Assessment of SARS-CoV-2-longterm morbidity and sequels on the population level:

In order to identify and treat these sequels in a timely fashion and to get a sense of the prevalence of such SARS-CoV-2 sequels on the population level, it is important to collect follow-up data and to comprehensively re-examine a population-representative sample of SARS-CoV-2 infected individuals.

Within the COVIDOM study we will conduct deep clinical and biochemical phenotyping in population-representative samples in Germany. This will allow novel insights into disease pathogenesis and chronicity of virus infections.

DETAILED DESCRIPTION:
Background:

COVID-19 is a novel disease caused by SARS-CoV-2. Severity of infection in the acute phase ranges from asymptomatic to critically ill and fatal courses of the disease. Besides the acute respiratory distress syndrome (ARDS), also thromboembolic events and acute damages of other organs are contributing to severe and critical courses of the disease in the acute phase of the infection.

It is, however, largely unknown whether and to what extent different organs are affected in individuals with milder courses of the disease.

Hypotheses:

1. Across all severity stages in the acute phase, SARS-CoV-2 infection causes longterm damages in various organ systems in a significant proportion of patients.
2. Beyond the damages directly caused by the infection, also the behavioral changes implemented to reduce the spread of the virus might impact an individual's health status and quality of life.
3. The infection itself and the pandemic in general results in increased use of health care resources.

Methods:

SARS-CoV-2 infected individuals in defined geographic regions will be contacted through the responsible health authorities and will be informed about the study and invited to participate. These individuals will presumably represent all severity grades in the initial phase of the infection (asymptomatic, uncomplicated, complicated, critical course of disease) and each of them will be offered a detailed clinical examination program that Includes structural and functional assessment of various organ systems (lungs, cardiovascular, CNS including smell/tase, liver), a comprehensive medical history, as well as psychological and psychiatric assessments.

ELIGIBILITY:
Inclusion Criteria:

* PCR-confirmed SARS-CoV-2 infection
* living in one of the target areas
* age at least 18 years
* written informed consent

Exclusion Criteria:

* Acute SARS-CoV-2 infection or reinfection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: SARS-CoV-2 infected individuals in defined geographic regions will be contacted through the responsible health authorities and will be informed about the study and invited to participate. These individuals will presumably represent all severity grades in the initial phase of the infection (asymptomatic, uncomplicated, complicated, critical course of disease) and each of them will be offered a detailed clinical examination program that Includes structural and functional assessment of various organ systems (lungs, cardiovascular, CNS including smell/tase, liver), a comprehensive medical history, as well as psychological and psychiatric assessments.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-11-16 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Longterm morbidities and sequels of SARS-CoV-2 infections in the general population | Preliminary results in 03/2021
  Chronic organ impairments, especially of the lungs, heart, liver, central nervous system, smell and taste or psychological well-being bases on functional assessments (i.e. lung function including forced spirometry, bodyplethysmography, diffusing capacity for CO, FeNO, echocardiography, testing of smell and taste, neurological assessment, psychological assessment) and biomarker studies (blood, nasopharyngeal swabs, urin, stool)

SECONDARY OUTCOMES:
Longterm quality of life of SARS-CoV-2 infected individuals recruited from the general population | Preliminary results in 03/2021
  Longitudinal assessment of general and health-related quality of Life, as well as health status in SARS-CoV-2 infected individuals of different severity grades
Longterm health care utilization of SARS-CoV-2 infected individuals recruited from the general population | Preliminary results in 03/2021
  Longitudinal assessment of health-care utilization based on insurance data in SARS-CoV-2 infected individuals of different severity grades

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Schreiber, Prof. Dr., Study Director — Internal Medicine Department I, UKSH Kiel
Locations (3):
- Germany (3):
  - University Hospital Wuerzburg, Würzburg, Bavaria
  - University Hospital Schleswig-Holstein, Campus Kiel, Kiel, Schleswig-Holstein
  - University Hospital Charité Berlin, Berlin

IPD SHARING:
Plan to Share IPD: No
Please see use and access conditions according to www.napkon.de

REFERENCES:
- [Derived] Appel KS, Lee CH, Nunes de Miranda SM, Maier D, Reese JP, Anton G, Bahmer T, Ballhausen S, Balzuweit B, Bellinghausen C, Blumentritt A, Brechtel M, Chaplinskaya-Sobol I, Erber J, Fiedler K, Geisler R, Heyder R, Illig T, Kohls M, Kollek J, Krist L, Lorbeer R, Miljukov O, Mitrov L, Nurnberger C, Pape C, Pley C, Schafer C, Schaller J, Schattschneider M, Scherer M, Schulze N, Stahl D, Stubbe HC, Tamminga T, Tebbe JJ, Vehreschild MJGT, Wiedmann S, Vehreschild JJ. A precise performance-based reimbursement model for the multi-centre NAPKON cohorts - development and evaluation. Sci Rep. 2024 Jun 13;14(1):13607. doi: 10.1038/s41598-024-63945-5. PMID 38871878
- [Derived] Hartung TJ, Bahmer T, Chaplinskaya-Sobol I, Deckert J, Endres M, Franzpotter K, Geritz J, Haeusler KG, Hein G, Heuschmann PU, Hopff SM, Horn A, Keil T, Krawczak M, Krist L, Lieb W, Maetzler C, Montellano FA, Morbach C, Neumann C, Nurnberger C, Russ AK, Schmidbauer L, Schmidt S, Schreiber S, Steigerwald F, Stork S, Zoller T, Maetzler W, Finke C; NAPKON Study Group. Predictors of non-recovery from fatigue and cognitive deficits after COVID-19: a prospective, longitudinal, population-based study. EClinicalMedicine. 2024 Feb 3;69:102456. doi: 10.1016/j.eclinm.2024.102456. eCollection 2024 Mar. PMID 38333368
- [Derived] Schons M, Pilgram L, Reese JP, Stecher M, Anton G, Appel KS, Bahmer T, Bartschke A, Bellinghausen C, Bernemann I, Brechtel M, Brinkmann F, Brunn C, Dhillon C, Fiessler C, Geisler R, Hamelmann E, Hansch S, Hanses F, Hanss S, Herold S, Heyder R, Hofmann AL, Hopff SM, Horn A, Jakob C, Jiru-Hillmann S, Keil T, Khodamoradi Y, Kohls M, Kraus M, Krefting D, Kunze S, Kurth F, Lieb W, Lippert LJ, Lorbeer R, Lorenz-Depiereux B, Maetzler C, Miljukov O, Nauck M, Pape D, Puntmann V, Reinke L, Rommele C, Rudolph S, Sass J, Schafer C, Schaller J, Schattschneider M, Scheer C, Scherer M, Schmidt S, Schmidt J, Seibel K, Stahl D, Steinbeis F, Stork S, Tauchert M, Tebbe JJ, Thibeault C, Toepfner N, Ungethum K, Vadasz I, Valentin H, Wiedmann S, Zoller T, Nagel E, Krawczak M, von Kalle C, Illig T, Schreiber S, Witzenrath M, Heuschmann P, Vehreschild JJ; NAPKON Research Group. The German National Pandemic Cohort Network (NAPKON): rationale, study design and baseline characteristics. Eur J Epidemiol. 2022 Aug;37(8):849-870. doi: 10.1007/s10654-022-00896-z. Epub 2022 Jul 29. PMID 35904671
- [Derived] Bahmer T, Borzikowsky C, Lieb W, Horn A, Krist L, Fricke J, Scheibenbogen C, Rabe KF, Maetzler W, Maetzler C, Laudien M, Frank D, Ballhausen S, Hermes A, Miljukov O, Haeusler KG, Mokhtari NEE, Witzenrath M, Vehreschild JJ, Krefting D, Pape D, Montellano FA, Kohls M, Morbach C, Stork S, Reese JP, Keil T, Heuschmann P, Krawczak M, Schreiber S; NAPKON study group. Severity, predictors and clinical correlates of Post-COVID syndrome (PCS) in Germany: A prospective, multi-centre, population-based cohort study. EClinicalMedicine. 2022 Jul 18;51:101549. doi: 10.1016/j.eclinm.2022.101549. eCollection 2022 Sep. PMID 35875815
- See also: Related Info — http://www.covidom.de
- See also: Related Info — http://www.napkon.de